CLINICAL TRIAL: NCT05345236
Title: A Phase III Randomised, Double-masked, Parallel Group Study to Compare the Efficacy and Safety Between QL1207 (Proposed Aflibercept Biosimilar) and Eylea® in Subjects With Wet Age-related Macular Degeneration
Brief Title: A Study to Compare QL1207 to Eylea® in Subjects With Wet Age-related Macular Degeneration (wAMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1207-002
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1207 (Experimental): Subjects randomized into QL1207 group will receive QL1207 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  Interventions: Drug: Aflibercept
- Eylea® (Active Comparator): Subjects randomized into Eylea® group will receive Eylea® 2 mg (0.05 mL) via intravitreal injection every 4 weeks for the first 3 months, followed by 2 mg (0.05 mL) once every 8 weeks until Week 48.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal (IVT) injection
  Other Names: Eylea， VEGF-Trap

SUMMARY:
This is a randomised, double-masked, parallel group, multicentre study to evaluate the efficacy and safety of QL1207 compared to Eylea® in subjects with wet AMD.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either QL1207 or Eylea® (administered via intravitreal [IVT] injection 2 mg [0.05 mL] every 4 weeks for the first 3 months (i.e., at Weeks 0, 4, and 8), followed by 2 mg [0.05 mL] once every 8 weeks ) . Subjects will be administered the study drug up to week 48, and the last assessment will be done at Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years male and female
2. Treatment naïve, *active subfoveal choroidal neovascularisation (CNV) lesion secondary to AMD in the study eye
3. CNV area ≥50% of total lesion size
4. Total lesion area ≤ 12.0 Disc Areas (DA) in size (including blood, scars, and neovascularisation) in the study eye
5. BCVA of 20/40 to 20/200 (letter score of 73 to 34, inclusive) using ETDRS charts in the study eye
6. Fellow eye is not expected to need any anti-VEGF treatment for the duration of study participation.

Exclusion Criteria:

Study eye:

1. Sub- or intra-retinal haemorrhage that comprises more than 50% of the entire lesion or presence of blood with the size of 1 DA or more involving the centre of fovea
2. Scar, fibrosis, or atrophy involving the centre of the fovea
3. Presence of CNV due to other causes, such as ocular histoplasmosis, trauma, multifocal choroiditis, angioid streaks, history of choroidal rupture, or pathologic myopia
4. Any concurrent macular abnormality other than AMD which could affect central vision or the efficacy of IP
5. Current vitreous haemorrhage within 30days before randomization
6. Any other intraocular surgery or periocular surgery within 90 days prior to randomisation, except for lid surgery, which may not have taken place within 30 days prior to randomisation.
7. Uncontrolled ocular hypertension (defined as intraocular pressure [IOP] ≥ 25 mmHg despite treatment with anti-glaucoma medication) at Screening

   Either eye:
8. Any previous IVT anti-vascular endothelial growth factor (VEGF) treatment
9. Any previous systemic anti-VEGF treatment
10. History of treatment involving macula such as macular laser photocoagulation, photodynamic therapy (PDT), transpupillary thermotherapy (TTT), radiation therapy, or any ocular treatment for neovascular AMD
11. Active or suspected ocular and periocular infection at Screening or at randomisation
12. History of idiopathic or autoimmune-associated uveitis

    Other:
13. Known allergic reactions and/or hypersensitivity to any component of Eylea or QL1207 or allergy to the fluorescein sodium for injection in angiography
14. Uncontrolled systemic hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 95 mmHg on optimal medical regimen)
15. Any previous systemic anti-VEGF treatment
16. Women of childbearing potential who are pregnant, planning to become pregnant, lactating, or not using adequate birth control, as specified in protocol. For women of childbearing potential, a serum pregnancy test must result negative at Screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) Change From Baseline (No. of Letters) to Week 12 | Baseline (Day 0), Week 12

SECONDARY OUTCOMES:
Proportion of subjects who gained at least 5,10 and 15 lettersbaseline to week 12,week 24 and week 52 | Baseline (Day 0), Week 12, Week 24, Week 52
Change From Baseline in CRT(central retina thickness) by visit | Baseline (Day 0), week 4, week 8, Week 12, Week 24, Week 52
BCVA Change From Baseline by visit | Baseline (Day 0), Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52
Change from baseline in CNV area from baseline to week 12, week 24 and week 52 | Baseline (Day 0), Week 12, Week 24, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: youxin chen, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li B, Fan K, Zhang T, Wu Z, Zeng S, Zhao M, Ren Q, Zheng D, Wang L, Liu X, Han M, Song Y, Ye J, Pei C, Yi J, Wang X, Peng H, Zhang H, Zhou Z, Liang X, Yu F, Wu M, Li C, Lei C, Hao J, Tang L, Yuan H, Cai S, Li Q, Zhong J, Li S, Liu L, Ke M, Wang J, Wang H, Zhu M, Wang Z, Yan Y, Wang F, Chen Y. Efficacy and Safety of Biosimilar QL1207 vs. the Reference Aflibercept for Patients with Neovascular Age-Related Macular Degeneration: A Randomized Phase 3 Trial. Ophthalmol Ther. 2024 Jan;13(1):353-366. doi: 10.1007/s40123-023-00836-4. Epub 2023 Nov 21. PMID 37987893